CLINICAL TRIAL: NCT02760381
Title: Acetic Acid for Optical Characterization of Colonic Polyps: A Feasibility Study
Brief Title: Acetic Acid for Optical Characterization of Colonic Polyps
Acronym: ATOMIC I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ATOMIC I
Record Dates: First submitted 2016-04-23; First posted 2016-05-03 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Routine colonoscopy Cohort (Experimental): Patients receiving routine colonoscopy receive the intervention: NBI + Acetic Acid (AA)
  Interventions: Device: NBI + Acetic Acid (AA)

INTERVENTIONS:
Device: NBI + Acetic Acid (AA) — Patients belonging to the Routine colonoscopy Cohort will receive NBI + Acetic Acid (AA) chromoendoscopy for optical predictions of colonic polyps.

SUMMARY:
Adenomas and hyperplastic polyps are polypoid lesions that can occur in any part of the colon. Currently all polyps should be resected endoscopically, however adenomas have the potential to develop into colorectal cancer whereas hyperplastic polyps do not. This approach enables the lesions to be evaluated under the microscope. Currently only the pathological diagnosis can distinguish exactly between adenomas and hyperplastic polyps. Acetic acid (AA) chromoendoscopy is already widely used in order to improve optical determination of mucosal lesions in the upper gastrointestinal tract. In the colon only few studies investigated the impact of AA in differentiating normal mucosa from suspicious mucosa. The aim of the present study is to evaluate the value of spraying acetic acid as an adjunct for optical characterization of colon polyps. Using AA may be beneficial for determining optical diagnoses of colon polyps during real time colonoscopy. This is a single-arm proof of principle study. If colon polyps are found during colonoscopy a 1.5 percent AA solution will be used for chromoendoscopy. Endoscopists are encouraged to use the Narrow Band Imaging (NBI) function of the endoscope prior to the use of AA. After AA is sprayed endoscopists will diagnose the polyp optically. Endoscopists have to predict adenomatous or non-adenomatous histology based upon optical features of the polyp. All polyps will be resected endoscopically so that histopathological diagnoses can be determined. After completing the trial the investigators aim to compare optical and histopathological-based diagnoses of polyps. Histopathological diagnoses will serve as the gold standard. Based upon this information the accuracy of the optical diagnoses will be calculated. The investigators hypothesis is, that optical-based diagnosis using NBI and AA will be accurate in > 75% of all polyp cases.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy

Exclusion Criteria:

* pregnant women
* emergency investigation
* history of inflammatory bowel disease
* contraindication for polyp resection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic test: Optical characterization of colon polyps | up to 2 weeks
  Optical diagnosis of polyp histology will be assessed within a period of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München München, Deutschland Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No